CLINICAL TRIAL: NCT07105891
Title: Optimization of Oocyte Warming Protocols: a Comparative Study of Standard, Rapid, and Ultra-rapid Techniques on Oocyte Survival Rate and Spindle Morphometry
Brief Title: Optimization of Oocyte Warming Protocols
Acronym: OVOfast
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Enrico Papaleo, MD, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OVOfast
Record Dates: First submitted 2025-06-19; First posted 2025-08-06 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Oocyte Cryopreservation
Keywords: oocytes; thawing; art; vitrification; warming; survival rates

STUDY DESIGN:
Intervention Model Description: sibling design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard (Other): Standard thawing
  Interventions: Other: Thawing protocol
- Fast (Other): Fast thawing
  Interventions: Other: thawing protocol
- Ultrafast (Other): Ultrafast thawing
  Interventions: Other: thawing protocol

INTERVENTIONS:
Other: Thawing protocol — Standard thwaing
  Arms: Standard
Other: thawing protocol — Fast thawing
  Arms: Fast
Other: thawing protocol — Ultrafast thawing
  Arms: Ultrafast

SUMMARY:
This is a retrospective study with a sibling design comparing new oocyte thawing protocols (rapid and ultra-rapid) with the traditional method

ELIGIBILITY:
Inclusion Criteria:

* Vitrified oocytes from the Centro Scienze della Natalità, IRCCS San Raffaele Hospital
* Patients who explicitly consented to the disposal of their stored gametes and authorized their use for research purposes through the informed consent process
* Oocytes cryopreserved using the vitrification technique
* Patients age 20-39 yo

Exclusion Criteria:

* All oocytes cryopreserved using the slow freezing technique
* Oocytes from patients older than 40 years

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 399 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Oocytes Survival rate | 2 hours post-warming
  Oocyte survival rate will be assessed 2 hours after thawing using morphological evaluation under a light microscope. Surviving oocytes will be identified by the presence of an intact zona pellucida and oolemma, a round shape, and homogeneous cytoplasm without signs of lysis, fragmentation, or cytoplasmic granulation.

SECONDARY OUTCOMES:
Spindle configuration | 2 hours post thawing
  Spindle configuration in thawed oocytes will be assessed using confocal microscopy following immunofluorescence staining. The spindles will be classified as normal, slightly aberrant, or aberrant.
Chromosome distribution | 2 hours post thawing
  Chromosome distribution will be assessed using confocal microscopy following immunofluorescence staining. The distribution will be classified as normal, misaligned, or displaced.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No